CLINICAL TRIAL: NCT06214949
Title: Personalized Repetitive Transcranial Magnetic Stimulation (PrTMS) as a Treatment for Chronic Neck Pain
Brief Title: Personalized Repetitive Transcranial Magnetic Stimulation (PrTMS)
Acronym: PrTMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-0324
Record Dates: First submitted 2023-12-19; First posted 2024-01-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Personalized Repetitive Transcranial Magnetic Stimulation (Experimental)
  Interventions: Device: Personalized Repetitive Transcranial Magnetic Stimulation
- Sham Personalized Repetitive Transcranial Magnetic Stimulation (Experimental)
  Interventions: Device: Sham Personalized Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Personalized Repetitive Transcranial Magnetic Stimulation — Treatment will consist of 15 sessions over 3-4 weeks. Specifically, the active or sham treatments will be conducted ~5 times a week during the treatment phase of the study. The treatment protocol parameters (stimulus location, frequency, duration, and intensity) will be derived from the PrTMS software algorithm which incorporates clinical inputs from neurocognitive surveys and quantitative EEG analysis. The mechanical parameters will adhere to the recommended PrTMS parameters for pain treatment: figure of 8 coil that produces biphasic stimulatory pulses to the central zone cortex, frontal zone cortex, Broca's area, and frontal pre-cortex areas at a stimulation depth of 2 cm. Treatment parameters will be unique to each participant but will remain within known ranges. The frequency will be between 8 and 13 Hz, at an amplitude of 20-30% (approximately 30-40% of RMT), and about 3200-7200 pulses per session. Since parameters are specific to each participant, treatment settings will vary.
  Arms: Personalized Repetitive Transcranial Magnetic Stimulation
Device: Sham Personalized Repetitive Transcranial Magnetic Stimulation — Treatment will consist of 15 sessions over the course of 3-4 weeks. More specifically, the active or sham treatments will be conducted roughly 5 times a week during the course of the treatment phase of the study. The TMS system will have three coils, one designated active and the other two unlabeled and identical in appearance, weight, and noises emitted, one of which will be active and one of which will be sham.
  Arms: Sham Personalized Repetitive Transcranial Magnetic Stimulation

SUMMARY:
This study aims to assess the efficacy of Personalized Repetitive Transcranial Magnetic Stimulation (PrTMS) therapy to reduce chronic neck for military health system beneficiaries.

DETAILED DESCRIPTION:
The objective of our proposed research is to (a) assess the efficacy of PrTMS therapy in reducing pain for military health system beneficiaries with chronic neck pain receiving standard of care* at Walter Reed National Military Medical Center, and (b) to describe participants' perceptions of PrTMS treatment and its perceived effect on their pain.

The specific aims for this study are as follows:

Specific Aims

Aim 1a: To assess the efficacy of PrTMS therapy in reducing pain for military health system beneficiaries with chronic neck pain receiving standard of care at Walter Reed National Military Medical Center.

Aim 1b: To describe participants' perceptions of PrTMS treatment and its perceived effect on their pain.

Hypothesis 1a: Participants receiving PrTMS therapy in addition to standard of care will report a significant mean reduction in their pain based on quantitative and qualitative assessments, when compared to standard of care plus sham PrTMS.

Hypothesis 1b: Participant response to PrTMS will be independent of patient demographics (age, race, sex), length of chronic pain, characterization of type of pain (e.g., sharp, burning, aching, etc.), or location of pain (e.g., local vs. radiating).

Outcome Measures:

DVPRS summary pain score and four supplemental questions, measuring activity, sleep, mood, and stress.

Aim 2: To examine the short- and intermediate-term changes in self-reported quality of life and biopsychosocial symptoms related to pain in military health system beneficiaries receiving PrTMS in addition to standard of care for chronic neck pain at Walter Reed National Military Medical Center.

Hypothesis 2: Participants receiving PrTMS therapy will report significantly lower mean scores on PROMIS (fatigue, pain interference, and social isolation) and sleep disturbance, and higher mean PROMIS (physical function and satisfaction with social roles) than participants receiving sham PrTMS across the intervention period and at follow up.

Outcome Measures:

The National Institutes of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) measures are validated, global measures of patient-reported outcomes with standardized scales and computer adaptive testing (CAT). CAT allows for reduced participant burden, as the number of questions asked to arrive at a score are fewer. PROMIS measures have also been recommended as an assessment tool for studies conducted exploring TMS as treatment for pain. To measure the biopsychosocial elements of pain, the following PROMIS measures will be utilized:

1. PROMIS Bank v1.0 - Fatigue
2. PROMIS Bank v1.1 - Pain Interference
3. PROMIS Bank v2.0 - Physical Function
4. PROMIS Bank v2.0 - Satisfaction with Social Roles
5. PROMIS Bank v1.0 - Social Isolation

Aim 3: To assess the impact that confounding factors such as depression, anxiety, sleep disorders, or PTSD may have on the efficacy of PrTMS as an augmentation to standard of care.

Hypothesis 3: Participants that have high premorbid levels of mental health disease or sleep disturbances will exhibit less response to PrTMS than those who do not.

Outcome Measures:

PCL-5, PHQ-9, SCI, GAD-7 and OURA ring. (see section 10.2)

Aim 4: To assess the short- and intermediate-term changes in plasma neuropeptides, inflammatory proteins and nucleic acids that can serve as blood based biomarkers for pain /stress.

Hypothesis 4: Participants receiving PrTMS therapy will demonstrate significantly lower mean plasma concentrations of tested plasma neuropeptides and inflammatory proteins, as well as associated genetic markers, including mRNA, miRNA, and genomic sequences.

Biological Blood and Serum Measures:

Neuropeptides such as ACTH, NPY, IGF-1, BDNF, NSE, GFAP, S100B; inflammatory proteins, such as IL-1beta, IL-2, IL-6, IL-8, IL-10, IL-12, TNF-alpha, IFN-gamma, MCP1/CCL2, CRP; mRNA; miRNA; and whole genome sequencing (WGS)

ELIGIBILITY:
Inclusion Criteria:

* Military health care beneficiary for enrollment.
* Over the age of 18 years.
* Presence of chronic neck pain for at least 3 months.

Exclusion Criteria:

* History of seizure, bipolar disorder, or schizophrenia.
* Unstable heart or pulmonary disease.
* Brain tumor, active brain infection, history of cerebral vascular accident (CVA), or penetrating brain injury.
* Use of medications that potentially lower seizure threshold without concomitant administration of anticonvulsant drugs that may protect against seizure occurrence.

  1. Antiviral medications and antipsychotic medications
  2. Recent withdrawal from sedatives
  3. Substance abuse of phencyclidine, amphetamines, ketamine, and gammahydroxybutyrate
* Not a suitable candidate for the study as determined by the PI.
* Pregnancy, breastfeeding, or plans to become pregnant during the course of the study.
* Presence of metallic hardware in close contact to the discharging coil (e.g. cochlear implants, internal pulse generator).
* Presence of implanted brain electrodes (cortical or deep-brain electrodes).
* Potential participants who score above a certain suicide relevant survey score on the Suicide Behaviors Questionnaire-Revised (SBQ-R), or are judged by expert clinicians to be a serious risk of harm to self, will be excluded.
* Participants cannot have undergone a previous TMS treatment within the last 30 days before the start of study treatment.
* Participants must have reliable and consistent access to the internet to complete surveys when not present in the clinic.
* Participants must not have a clinical diagnosis of insomnia.
* Participants can not be actively partaking in a substance abuse program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Defense & Veterans Pain Rating Scale (DVPRS) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements taken everyday during Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The DVPRS was developed to standardize pain measurement across all health care settings and promote pain assessment and reassessment practices. DVPRS is a visual pain scale to assess individual's pain intensity on a scale of 0-10, with an additional 4 questions to assess pain's interference with the participant's activity, sleep, mood, and stress. The scale has excellent internal reliability and test-retest reliability.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The PGIC outcome measure evaluates a patient's self-reported level of pain and their feelings about treatment effectiveness to determine symptom improvement using a 7 point scale from 1-7. Higher scores indicate a greater improvement while lower scores indicate less improvement or even worsening of a condition.
TMS Tolerability Worksheet (TTW) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The TTW is administered after each PrTMS session to accurately track and record tolerability of TMS therapy as well as frequency and severity of the known minor negative side effects of TMS, such as headaches.
Pain Anxiety Symptom Scale Short Form 20 (PASS) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The PASS measures anxiety and fear specifically related to pain on a scale from 0 (never) to 5 (always).
Sleep Condition Indicator (SCI) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The SCI is an 8-item self-report measure that evaluates insomnia disorder where answers to a given item are weighted from 0 (affected sleep) to 4 (no affected sleep). A higher score is indicative of better sleep.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The GAD-7 is a 7-item self-report measure that assesses an individual's level of anxiety on daily life using a scale from 0 (Not at all) to 3 (Nearly every day). Higher scores indicate higher levels of anxiety.
Patient Health Questionnaire (PHQ-9) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The (PHQ-9) is a 9-item measure of depression through affect on everyday life on a scale of 0 (Not at all) to 3 (Nearly every day). Higher scores are indicative of higher levels of depression.
Quantitative Analgesic Questionnaire (QAQ) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The QAQ is a tool used to identify and comprehensively document medication use and adherence to prescriptions based on patient self-reports.
Suicide Behaviors Questionnaire-Revised (SBQ-R) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The SBQ-R is a self-report questionnaire targeted to assess suicidal risk factors in individuals aged 13 and older. Responses will be scored based on how participants respond with values between 1 and 6 points. Higher scores are more indicative of suicidal risk.
PTSD Checklist for DSM-5 (PCL-5) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The PCL-5 is a self-report questionnaire on the presence and severity of PTSD symptoms. Responses range from values of 0 (Not at all) to 4 (Extremely) where higher scores are more indicative of severe PTSD.
Patient Reported Outcomes Measurement Information System (PROMIS) Scales. | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The PROMIS scales will be used in this study to examine effects of TMS on quality of life using the following scales: Fatigue, Pain Interference, Physical Function, Satisfaction with Social Roles, and Social Isolation. Responses will vary from Never (scored as 0) to Always (scored as 4). Higher scores being more indicative of the concept being measured.
Pittsburgh Sleep Quality Index (PSQI) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The PSQ-I is an effective instrument used to measure the quality and patterns of sleep in adults. Responses to questions about sleep will be scored from 0 (better sleep quality) to 3 (worse sleep quality). Higher overall scores being indicative of lower quality of sleep.
Insomnia Severity Index (ISI) | Measured to compare changes from Baseline; during Phase 1 and 2 of treatment; and during the follow up phase after treatment ends up to 8 weeks. Measurements will be taken once at end of Baseline, Phase 1 and Phase 2 and at 2, 4, and 8 weeks in Follow-Up
  The ISI is a 7-item measure designed to briefly assess the severity of both nighttime and daytime insomnia symptoms. Responses will vary from Not at all (scored as 0) to Very Much (score as 4). Higher scores being indicative of increasing level of insomnia.
Demographics Survey | Taken at Baseline to create comparable groups of treatment and will be used as covariates in statistical analysis.
  Demographics and Health Questionnaires has questions pertinent to this research effort, including: age, sex, relationship status, race/ethnicity, education, military service, deployment history, health history, current and prior treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseyi Gbade-Alabi, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States